CLINICAL TRIAL: NCT06772961
Title: Effect of Percutaneous Electrical Acupoint Stimulation on the Improvement of Incidence of Adverse Respiratory Events in the Emergence Period From General Anesthesia After Tracheal Extubation: A Single-center Randomized Controlled Study
Brief Title: Effect of Percutaneous Electrical Acupoint Stimulation on the Improvement of Incidence of Adverse Respiratory Events
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20240613-06-KS-01
Record Dates: First submitted 2025-01-01; First posted 2025-01-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Extubation; Respiratory Depression; Acupuncture Points; Hypoxia
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEAS group (Experimental): Transcutaneous electrical acupoint stimulation (TEAS) merges transcutaneous electrical nerve stimulation with acupoint therapy. It has its roots in acupuncture and shares similar effects, while being distinguished by its simplicity, safety, non-invasiveness, and reduced complications. TEAS functions by stimulating nerve fiber endings, which generates action potentials that are transmitted to the spinal cord and brain, subsequently triggering the release of related chemical mediators and producing corresponding physiological effects.
  In this study, the traditional acupoints Taiyuan on the lung meridian and Hegu on the large intestine meridian were selected. The lung and large intestine meridians are interconnected, so the combined application of Taiyuan and Hegu acupoints with TEAS can produce a synergistic effect. This combination enhances the replenishment of lung qi, promotes the flow of meridians, regulates qi, and disseminates lung functions. It can stimulate effective
  Interventions: Other: Transcutaneous electrical acupoint stimulation
- Control group (Placebo Comparator): conventional care plan
  Interventions: Other: Conventional care plan

INTERVENTIONS:
Other: Transcutaneous electrical acupoint stimulation — In this study, the traditional acupoints Taiyuan (LU9) on the lung meridian and Hegu (LI4) on the large intestine meridian were selected. The lung and large intestine meridians are interconnected, so the combined application of Taiyuan and Hegu acupoints with TEAS can produce a synergistic effect. This combination enhances the replenishment of lung qi, promotes the flow of meridians, regulates qi, and disseminates lung functions. It can stimulate effective breathing in patients, thus positively influencing the improvement of their oxygen saturation levels.
  Arms: TEAS group
Other: Conventional care plan — Conventional care plan
  Arms: Control group

SUMMARY:
The goal of this study is to investigate the effect of combined acupoint electrical stimulation at Taiyuan (LU9) and Hegu (LI4) on improving the incidence of respiratory adverse events after extubation in patients during the recovery period from general anesthesia.

The main content of this study involves selecting patients who have undergone general anesthesia and are admitted to the Post Anesthesia Care Unit (PACU), with an expected 236 participants. The researchers will randomly assign participants to either the TEAS group or the control group using a random number table. In the TEAS group, electrodes will be applied to the upper limbs at the Taiyuan and Hegu acupoints, without intravenous infusion, and connected to a stimulation device. The stimulation will use a frequency of 2/100 Hz with sparse-dense waves, and the intensity will be adjusted to the maximum current that the patient can tolerate, starting at the time of extubation and continuing for 30 minutes. The control group will receive routine care. Throughout the process, no invasive procedures will be performed.

In the PACU, the participants will:

Be positioned in a 30° head-up tilt position, with continuous ECG monitoring. The SpO2 alarm on the monitor will be set to 95%.

The same anesthesiologist will perform extubation according to the extubation criteria.

After extubation, participants will receive routine oxygen therapy via a nasal cannula at 3L/min with a CO2 end-expiratory monitoring module attached to the other end of the cannula. Simultaneously, the TEAS group will undergo transcutaneous electrical stimulation for 30 minutes, or the control group will receive routine care.

Participants will be observed in the PACU for at least 30 minutes. If no adverse events occur and the Steward score is ≥4, the patient will be deemed ready for discharge and escorted back to the ward. If there is any significant change in the patient's condition, they will be transferred to the ICU .

If any respiratory-related adverse events occur, measures such as awakening the patient, supporting the jaw, increasing oxygen flow, or administering mask oxygen will be taken to ensure patient safety, and these events will be recorded in the "PACU Postoperative General Anesthesia Patient Condition Observation and Nursing Record."

DETAILED DESCRIPTION:
According to domestic and international studies, apnea, respiratory depression, desaturation, hypoxemia, and severe hypoxia are documented as adverse respiratory events during the recovery period. The post-anesthesia recovery phase is a high-risk period for hypoxemia. A brief decrease in SpO2 may indicate the onset of respiratory adverse events such as hypoxemia and severe hypoxia. Patients in the Post Anesthesia Care Unit (PACU) are in the early stages of awakening from general anesthesia, where their spontaneous breathing function gradually recovers. However, some patients may still experience residual effects of muscle relaxants or analgesics that lead to respiratory depression. After the removal of mechanical ventilation, patients often experience a decrease in SpO2. In an analysis by Wu Qiao et al. on the incidence of respiratory adverse events during the recovery period after extubation in gastrointestinal oncology patients under general anesthesia, the incidence of apnea was 50.85%, and respiratory depression occurred in 42.8% of cases. Notably, extubation in the PACU after general anesthesia marks a critical point in the transition from assisted to spontaneous breathing. Therefore, the incidence of respiratory adverse events in the early post-extubation period in the PACU is high. Desaturation, hypoxemia, and severe hypoxia in many patients are secondary to apnea or respiratory depression, and if not intervened in time, hypoxemia can occur and potentially endanger the patient's life. Hence, how to effectively reduce the incidence of respiratory adverse events in patients after general anesthesia extubation has become a focus of research in both academic and clinical practice.

Moreover, as China's aging population grows and medical technology continues to advance, the number of patients at risk for post-anesthesia hypoxemia is increasing. In the face of a significant rise in the workload of post-anesthesia recovery rooms, the capacity of PACU medical staff to anticipate and manage respiratory adverse events has not yet met clinical demands.

Transcutaneous electrical acupoint stimulation (TEAS) merges transcutaneous electrical nerve stimulation with acupoint therapy. Rooted in acupuncture, it offers similar effects and is characterized by its simplicity, safety, non-invasiveness, and fewer complications. TEAS functions by stimulating nerve fiber endings to generate action potentials, which are then transmitted to the spinal cord and brain, leading to the release of related chemical mediators and producing corresponding physiological effects. This study selected the primary acupoint Taiyuan (LU9) on the lung meridian and Hegu (LI4) on the large intestine meridian. The lung and large intestine meridians are interconnected, and the combined use of Taiyuan and Hegu acupoints with TEAS can have a synergistic effect, enhancing the replenishment of lung qi, promoting the flow of meridians, regulating qi, and disseminating lung functions. It can effectively stimulate patients' breathing, thereby improving oxygen saturation. However, there are currently few prospective studies on the role of TEAS with Taiyuan and Hegu in reducing the incidence of respiratory adverse events after extubation in patients during the recovery period of general anesthesia, and further in-depth exploration is needed.

Therefore, this study will employ the combined acupoint TEAS stimulation of Taiyuan and Hegu as an intervention method, aiming to explore its role in improving the incidence of respiratory adverse events after extubation in patients during the post-anesthesia recovery period. The goal is to provide more reliable scientific evidence for clinical practice. This study aims to offer new theoretical support for the nursing care of patients after extubation during the post-anesthesia recovery period and provide new ideas and methods for further improving patients' quality of life and surgical treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1: Age >18 years old.

  2: ASA I-III

  3: Patients undergoing elective general anesthesia surgery who are extubated upon arrival to the PACU

Exclusion Criteria:

* 1: Preoperative comorbidities include severe cardiovascular or respiratory diseases

  2: Serious reflux aspiration during the perioperative period

  3: Concurrent psychiatric disorders

  4: Local skin infections or nerve damage at the upper limb Taiyuan and Hegu acupoints

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Respiratory adverse events | After the patient enters the PACU from general anesthesia
  In this study, the respiratory status of patients was monitored using PetCO2 in conjunction with SpO2, and adverse respiratory events such as apnea, respiratory depression, desaturation, hypoxemia, and severe hypoxia were recorded during the recovery period of general anesthesia. Based on other studies, apnea in this study is defined as the cessation of the end-tidal CO2 waveform for a duration exceeding 20-30 seconds; respiratory depression is characterized by a respiratory rate of ≤5 breaths per minute, PetCO2 ≤15mmHg (1mmHg=0.133kPa) or ≥55mmHg, a change of ≥10mmHg from the baseline, or the absence of the end-tidal CO2 waveform for ≥30 seconds; desaturation refers to a decrease in SpO2, specifically when SpO2 drops to a range of 95% to 90% and persists for over 15 seconds; hypoxemia is indicated by an arterial oxygen partial pressure below 60mmHg or when SpO2 is between 90% and 85%; and severe hypoxia is defined as SpO2 falling below 85%.

SECONDARY OUTCOMES:
General adverse events other than hypoxia | After the patient enters the PACU from general anesthesia
  Including vomiting, regurgitation, aspiration, bronchospasm, choking,

OTHER OUTCOMES:
Adverse events related to transcutaneous electrical stimulation | After the patient enters the PACU from general anesthesia
  Skin allergy and local muscle spasm at the electrode attachment site

CONTACTS AND LOCATIONS:
Overall Officials: xiaoliang wang, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
In order to protect the privacy of participants, researchers decided not to make the data public. To obtain relevant data, researchers can be contacted if necessary.